CLINICAL TRIAL: NCT00790582
Title: A Multi-Center Controlled Screening Trial of Safety and Efficacy of Lithium Carbonate in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Acronym: Lithium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forbes Norris MDA/ALS Research Center (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Dr. Robert Miller, Director, Forbes Norris MDA/ALS Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28.013
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig's Disease; Lithium; Lithium Carbonate
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lithium carbonate (Experimental)
  Interventions: Drug: lithium carbonate

INTERVENTIONS:
Drug: lithium carbonate — The dosage of lithium carbonate will be adjusted for each individual. The maximum dose is 450mg/day.

SUMMARY:
This is a Phase II screening study of lithium carbonate in ALS. The purpose of this study is to find out if lithium carbonate is safe to be used in people with ALS and if it can slow the progression of the disease. Since there is no placebo in this study, all patients will be taking lithium carbonate.

DETAILED DESCRIPTION:
This is a Phase II Screening study. There is no placebo (inactive or 'fake' drug) in this study, meaning that all participants will be taking lithium carbonate. The purpose of this study is to find out if lithium carbonate is safe to be used in people with ALS and if it can slow the progression of the disease.

A recent article was published in a highly regarded medical journal that showed a positive effect of lithium carbonate on an ALS type mouse. The researchers then studied a very small number of people with ALS, giving 16 people lithium carbonate with riluzole and giving 28 people only riluzole. The people who took lithium remained stronger for a considerably longer period of time. However, the study was very small and we cannot really tell if lithium works unless a larger study is performed. It is not well understood why lithium carbonate might be helpful but it is believed that it may play a role in protecting the motor nerves from the damage of ALS.

If you choose to participate, you will need to go to your study clinic for research study visits 7 times in one year and you will have 4 telephone interviews during that time. These visits and phone calls could take up to 17 hours in total.

Caution: Lithium is an FDA approved drug used for some psychiatric disorders. It is not FDA approved for ALS. Lithium has many potentially serious side effects and must only be taken under close supervision of your physician.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of laboratory-supported probable, probable, or definite ALS
* Vital capacity of at least 75% of predicted
* Onset of weakness within 3 years prior to enrollment
* If patients are on riluzole, they must be on a stable dose for at least 30 days prior to baseline visit
* Women of childbearing potential must be surgically sterile or using an effective method of birth control and have a negative pregnancy test
* Willing and able to give informed consent

Exclusion Criteria:

* Diagnosis of other neurodegenerative disease
* Need tracheotomy ventilation or non-invasive ventilation 23 or more hours/day
* Clinically significant history of any unstable medical condition in past 30 days
* History of renal
* History of liver disease
* Current pregnancy or lactation
* Use of lithium within thirty days of enrollment
* Significantly limited mental capacity
* History of recent drug or alcohol abuse
* Use of any investigational drug within 30 days prior to enrollment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Miller, MD, Study Director — California Pacific Medical Center
Locations (10):
- United States (10):
  - Mayo Clinic, Scottsdale, Arizona
  - UCLA Neuromuscular Research Center, Los Angeles, California
  - UC Irvine MDA/ALS & Neuromuscular Center, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Kansas University Medical Center, Kansas City, Kansas
  - Washington University Department of Neurology, St Louis, Missouri
  - Providence ALS Clinic, Portland, Oregon
  - University of Pennsylvania Neurological Institute, Philadelphia, Pennsylvania
  - Methodist Neurological Institute, Houston, Texas
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah

REFERENCES:
- [Background] Fornai F, Longone P, Cafaro L, Kastsiuchenka O, Ferrucci M, Manca ML, Lazzeri G, Spalloni A, Bellio N, Lenzi P, Modugno N, Siciliano G, Isidoro C, Murri L, Ruggieri S, Paparelli A. Lithium delays progression of amyotrophic lateral sclerosis. Proc Natl Acad Sci U S A. 2008 Feb 12;105(6):2052-7. doi: 10.1073/pnas.0708022105. Epub 2008 Feb 4. PMID 18250315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between May 2008 and February 2009. Inclusion criteria were a diagnosis of probable or definite ALS (12), age 21-85 years, forced vital capacity (FVC) greater than or equal to 75% of predicted, and onset of weakness within 3 years. Patients taking riluzole were on a stable dose for at least 30 days.
Pre-assignment Details: This was an open label single-arm Phase II screening trail. All enrolled subjects (n=109) were treated. Their results were compared with placebo subjects from an historical database of ALS placebo patients from recent studies (n=249). Thus the number enrolled (n=109) does not equal the total number of subjects (n=358).
  Enrolled subjects started lithium carbonate at 150 mg twice daily. If subjects did not tolerate a dose it was tapered by 150 mg increments to the maximum tolerated dosage.
Groups:
- Treatment: 109 subjects were assigned to treatment with lithium carbonate
- Control: 249 placebo subjects from previous clinical trials
Period: Overall Study
Arm/Group | Treatment | Control
Started | 109 | 249
Completed | 78 | 162
Not Completed | 31 | 87
Not completed — Death | 14 | 32
Not completed — Physician Decision | 7 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 7 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium Carbonate | Historical Controls | Total
Number analyzed (Participants) | 109 | 249 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.7) | 57.6 (11.0) | 57.2 (11.2)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 186 | 270
  >=65 years | 25 | 63 | 88
  18 to 75 years | 109 | 249 | 358
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 83 | 121
  Male | 71 | 166 | 237
Region of Enrollment [Number; unit: participants]
  United States | 109 | 249 | 358

OUTCOME MEASURES:

1. Primary Outcome: Change in Monthly Rate of Decline in ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Score - Revised)
Description: This questionnaire has 12 questions about the patient's ability to complete certain daily activities. There are three questions each about the mouth area, arms, legs, and breathing. A normal score is 48 with each question scored at 0 (worst) to 4 (normal function). In research studies, the change in slope is measured in number of points changed per month. Maximum possible=48 (normal) Minimum=0 (severe dysfunction)
Time Frame: Baseline, Month 1,3,4.5,6,7.5,9,10.5,12,13
Measure: Mean (95% Confidence Interval); unit: points per month
Arm/Group | Lithium Carbonate | Historical Controls
Number analyzed (Participants) | 109 | 249
points per month | 1.20 [1.04 to 1.35] | 1.01 [0.90 to 1.11]

2. Secondary Outcome: Vital Capacity
Description: Vital Capacity (VC) is a breathing test in which the patient is asked to take a deep breath and then blow out all of the breath through a tube. The volume is measured in number of liters. It is converted to a percent predicted for the patient's age, height, and gender.
Time Frame: Screen, Baseline, Month 1,3,6,9,12
Measure: Mean (95% Confidence Interval); unit: Decline in the percent predicted/month
Groups:
- Lithium Carbonate: Treatment arm
- Control: Placebo arm
Arm/Group | Lithium Carbonate | Control
Number analyzed (Participants) | 109 | 249
Decline in the percent predicted/month | 2.84 [2.36 to 3.32] | 2.91 [2.59 to 3.23]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for the duration of the trial (1 year).
Groups:
- Lithium Carbonate: Treated Patients
- Historical Controls: Placebo Patients
Arm/Group | Lithium Carbonate | Historical Controls
All-Cause Mortality (participants affected / at risk) | 14/109 | 44/249
Serious Adverse Events (participants affected / at risk) | 62/109 | 91/249
Other Adverse Events (participants affected / at risk) | 99/109 | 175/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=109) | Historical Controls (N=249)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 51 (51)
Gastrointestinal (Gastrointestinal disorders) | 17 (17) | 23 (23)
Other (General disorders) | 20 (20) | 17 (17)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=109) | Historical Controls (N=249)
Gastrointestinal (Gastrointestinal disorders) | 16 | 138 (406)
Cardiovascular (Cardiac disorders) | 1 | 46 (63)
Dermatological (Skin and subcutaneous tissue disorders) | 5 | 99 (211)
Ears, Nose, Throat (Ear and labyrinth disorders) | 6 | 86 (151)
Endocrine/Metabolic (Endocrine disorders) | 4 | 8 (8)
Genitourinary (Reproductive system and breast disorders) | 2 | 64 (109)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 | 85 (170)
Neurological (Nervous system disorders) | 27 | 98 (209)
Other (General disorders) | 4 | 7 (8)
Falls (Nervous system disorders) | 12 | 72 (194)
Psychological (Psychiatric disorders) | 4 | 56 (83)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 12 | 76 (123)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No